CLINICAL TRIAL: NCT02979015
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Single-Dose Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneously Administered Alirocumab in Chinese Healthy Subjects
Brief Title: A Study of Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous (SC) Administered Alirocumab in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PKD13404; U1111-1133-7871 (Other: UTN)
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alirocumab (Experimental): Subcutaneous injection of a single dose of alirocumab, dose level according to ascending dose design
  Interventions: Drug: alirocumab SAR236553 (REGN727)
- Placebo (Placebo Comparator): Subcutaneous injection of a single dose of matching placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: alirocumab SAR236553 (REGN727) — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous
  Arms: Alirocumab
Drug: placebo — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous
  Arms: Placebo

SUMMARY:
Primary Objective:

To assess the safety and tolerability of ascending single SC doses of alirocumab in Chinese healthy subjects.

Secondary Objectives:

* To assess the pharmacokinetic profile of a single SC dose of alirocumab.
* To assess the pharmacodynamic effect of a single SC dose of alirocumab on low-density lipoprotein cholesterol (LDL-C) and other lipid parameters.
* To assess the immunogenicity of a single SC dose of alirocumab.

DETAILED DESCRIPTION:
Ascending dose design includes 3 dose levels. Tolerance data up to at least 14 days post dosing from at least 6 subjects of the previous cohort will be reviewed before proceeding with a next dose. Total duration of the study per subject is approximately 15 weeks (including screening period).

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female subjects.
* Aged 18 to 45 years old.
* Low-density lipoprotein cholesterol >100 mg/dL (2.59 mmol/L).

Exclusion criteria:

* Subjects with any history or presence of clinically relevant illness.
* Serum triglycerides >200 mg/dL (2.26 mmol/L) measured after at least 10 hour fasting.
* Use of a medication or nutraceutical in order to alter serum lipids within 4 weeks prior to screening, including but not limited to statins, ezetimibe, fibrates, niacin, or bile acid resins. Use of probucol within 8 weeks prior to screening.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-11-29; Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events based on standard and systematic assessment including physical examinations, 12 lead ECGs, vital signs and laboratory tests | Up to 12 weeks
Incidence of injection site reactions | Up to 4 days

SECONDARY OUTCOMES:
Change from baseline in LDL-C | Up to 12 weeks
Change from baseline in other lipid parameters | Up to 12 weeks
Pharmacokinetics: Assessment of serum concentrations of alirocumab | Up to 12 weeks
Pharmacokinetics: Assessment of serum concentrations of PCSK9 | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 156001, Beijing, China

REFERENCES:
- [Derived] Li H, Wei Y, Yang Z, Zhang S, Xu X, Shuai M, Vitse O, Wu Y, Baccara-Dinet MT, Zhang Y, Li J. Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Alirocumab in Healthy Chinese Subjects: A Randomized, Double-Blind, Placebo-Controlled, Ascending Single-Dose Study. Am J Cardiovasc Drugs. 2020 Oct;20(5):489-503. doi: 10.1007/s40256-020-00394-1. PMID 32080823